CLINICAL TRIAL: NCT01912872
Title: Multicentric, Open-label, Randomized, Parallel--group Study to Evaluate the Efficacy and Safety of Omalizumab in a 12- Month Period, in Patients With Severe IgE-mediated Asthma Inadequately Controlled With High Doses of Corticosteroids.
Brief Title: Study to Assess the Efficacy and Safety of Omalizumab Treatment on ICS Reduction for Severe IgE-mediated Asthma
Acronym: MEXIC
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Termination was due to identified errors in data management handling after an internal audit by the sponsor performed by third party.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIGE025AMX02
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Severe IgE-mediated Asthma
MeSH Terms: interventions — Omalizumab; Budesonide; Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omalizumab + budesonide and formoterol (Experimental): Participants will receive Omalizumab every 2 or 4 weeks depending on IgE level and body weight and will also receive budesonide and formoterol according to maximum daily dose.
  Interventions: Drug: Omalizumab; Drug: Budesonide; Drug: Formoterol
- Budesonide and formoterol (Active Comparator): Participants will receive budesonide and formoterol according to maximum daily dose.
  Interventions: Drug: Budesonide; Drug: Formoterol

INTERVENTIONS:
Drug: Omalizumab — Subcutaneous injection dose according to the IgE level and body weight.
  Arms: Omalizumab + budesonide and formoterol
Drug: Budesonide — Budesonide (400 μg, 200 μg or 100 μg) tablets taken orally according to maximum daily dose.
Drug: Formoterol — Formoterol 12ug tablets taken orally according to maximum daily dose.
Drug: Budesonide — Budesonide (400 μg, 200 μg or 100 μg). Patients were instructed to take the inhaled budesonide doses every 12 hours following the specific administration instructions as per the manufactures' prescription information.
Drug: Formoterol — Formoterol 12ug. Patients were instructed to take the inhaled formoterol doses every 12 hours following the specific administration instructions as per the manufactures' prescription information.
  Arms: Budesonide and formoterol

SUMMARY:
Assess efficacy and safety of omalizumab treatment during 12 months in order to reduce the use of inhaled corticosteroid (ICS) in pediatric and adult participants with severe Immunoglobulin E (IgE)-mediated asthma inadequately controlled with high doses of corticosteroids.

DETAILED DESCRIPTION:
This was a multicentric, open label, randomized, parallel-group study with a 12-month treatment period. Participants were assigned to one of the 2 treatment groups, omalizumab plus budesonide/formoterol or budesonide/formoterol alone.

The study comprised 4 phases:

During the 4-week run-in phase adult participants received budesonide 800 mg and formoterol 24 mg. If a participant complied with all inclusion and exclusion criteria and had received the according-to-age run-in proposed doses during the last month, the participant continued to the stable-steroid phase.

During the 16-week stable-steroid phase, adult and pediatric eligible participants were randomized to one of the two treatment groups.

During the 8-week steroid-reduction phase, adult and pediatric participants reduced 25% of the budesonide baseline dose every 2 weeks, depending of the asthma control, until they reached a 100% reduction of the baseline dose. The clinical control of asthma was defined according to criteria (GINA 2012).

ELIGIBILITY:
Inclusion Criteria

* Male and female between 6 and 55 years old. If female, participant of childbearing potential must use a safe and efficacious birth control method.
* Asthma is considered as not well-controlled if participant has 3 or more of the following conditions:

  1. Persistent day symptoms with current therapy twice at week or more, (siblings, dyspnea, cough, chest pain, thoracic oppression).
  2. One or more night-time awakenings over the last 4 weeks.
  3. Any limitation of age-appropriated habitual activities.
  4. Need of rescue medication (short acting β2 agonist) for two or more occasions per week during the last 4 weeks before screening and 2 consecutive weeks within the 4 weeks before selection.
  5. Peak expiratory flow (PEF) or VEF1 <80% predicted or personal best (if known) this is not mandatory for pediatric participants (under 18 years old).
* Despite continuous treatment with high-dose inhaled corticosteroids (ICS) or oral corticosteroids (OCS) (CSO≥ 1 mg/kg/day) with or without controllers (As per GINA 2012 definition), the subject is receiving high doses of ICS (budesonide or its equivalent) and a long-acting β2-agonists(LABA) (formoterol) for the past 12 weeks at visit 0.
* At last one documented asthma exacerbation (defined as increase asthma symptoms requiring systemic corticosteroid rescue therapy) that requires visits to the emergency room or to be hospitalized in the past 12 months. It is also considered asthma exacerbation a non-planned visit that required rescue medication (β2-agonists and/or steroid nebulization every 20 minutes or β2-agonists inhaler shots every 20 minutes).
* Positive skin test or in vitro reactivity to a perennial aeroallergen, documented during the 12 months previous screening.
* IgE total concentration ranging from 30 to 1500 UI/ml.
* Body weight between 20 to 150 kg Exclusion Criteria
* Pregnant or lactating female or without safe and efficacious birth control method if of childbearing potential.
* Currently smokers or history of smoking 10 or more packs per year.
* Ex-smokers with a history of more than 10 years of smoking. As an exception, a participant with this criterion will be considered as eligible if the FEV1 reversibility of the first spirometry reaches 12%.
* Active lung disease other than asthma.
* Use of methotrexate, gold salts, troleandomycin, cyclosporine, immunosuppressants, gammaglobulin or any other type of monoclonal antibody used during the 6 months prior to the initial visit.
* Use of omalizumab during the 4 months prior to de screening visit.
* History of renal disease, cardiovascular disease, metabolic disease, hematologic disease, gastrointestinal disease, as well as immunodeficiency or cerebrovascular disease currently under treatment but not-controlled.
* History of hepatic, neurologic, oncologic or autoimmune disease.
* Participant under suspicion of having cancer.
* Participants with history of hypersensitivity to sucrose, histidine, polysorbate 20 as well as to monoclonal antibodies or gammaglobulin.
* Hypersensitivity to omalizumab or its excipients.
* Abnormal values of the blood chemistry laboratory tests, over 2 times the upper limit normal, that are considered clinically significant.
* Underage participant or any participant under vulnerable conditions who does not live with their parents or legal guardian.

Ages: 6 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 112 (Actual)
Dates: Start 2013-11-11 (Actual); Primary Completion 2015-08-06 (Actual); Study Completion 2016-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- Mexico (10):
  - Novartis Investigative Site, Tuxtla Gutiérrez, Chiapas
  - Novartis Investigative Site, México, Edo. de México
  - Novartis Investigative Site, Pachuca, Hidalgo
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Guadaljara, Jalisco
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Tepic, Nayarit
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, Nezahualcóyotl, State of Mexico
  - Novartis Investigative Site, Mérida, Yucatán

RESULTS

PARTICIPANT FLOW:
Groups:
- Pediatric Patients: Omalizumab + Budesonide and Formoterol: Participants received omalizumab injection for s.c. use 2 or 4 weeks according to the IgE level and body weight and budesonide + formoterol administered through an inhaler device.
- Pediatric Patients: Budesonide and Formoterol: Participants received budesonide + formoterol administered through an inhaler device.
- Adult Patients: Omalizumab + Budesonide and Formoterol: Participants received Omalizumab every 2 or 4 weeks as a subcutaneous injection dose according to the IgE level and body weight. Participants also received and budesonide + formoterol administered through an inhaler device.
- Adult Patients: Budesonide and Formoterol: Participants receive budesonide + formoterol administered through an inhaler device.
Period: Overall Study
Arm/Group | Pediatric Patients: Omalizumab + Budesonide and Formoterol | Pediatric Patients: Budesonide and Formoterol | Adult Patients: Omalizumab + Budesonide and Formoterol | Adult Patients: Budesonide and Formoterol
Started | 16 | 17 | 40 | 39
Completed Study Treatment at Month 12 | 11 | 13 | 30 | 27
Discontinued Treatment Prior to Month 12 | 5 | 4 | 10 | 11
Completed | 11 | 13 | 30 | 27
Not Completed | 5 | 4 | 10 | 12
Not completed — Lost to Follow-up | 2 | 3 | 5 | 5
Not completed — Other unspecified | 3 | 1 | 3 | 0
Not completed — Informed consent withdrawn | 0 | 0 | 1 | 1
Not completed — Non-compliance with lab inc/exclusion | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Unsatisfactory therapeutic effect | 0 | 0 | 0 | 2
Not completed — Withdrawal of study medication | 0 | 0 | 0 | 2
Not completed — Missing | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) population included participants who received at least one dose of study drug and had at least one post-baseline assessment of the primary or secondary efficacy variables.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pediatric Patients: Omalizumab + Budesonide and Formoterol | Pediatric Patients: Budesonide and Formoterol | Adult Patients: Omalizumab + Budesonide and Formoterol | Adult Patients: Budesonide and Formoterol | Total
Number analyzed (Participants) | 16 | 17 | 40 | 39 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.1 (3.32) | 12.4 (1.80) | 37.6 (10.01) | 38.7 (10.30) | 30.4 (14.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 28 | 28 | 70
  Male | 10 | 9 | 12 | 11 | 42

OUTCOME MEASURES:

1. Primary Outcome: The Mean Prescribed Budesonide Dose (μg) at Baseline
Description: prescribed budesonide dose (in μg) at Baseline in intention to treat population and in intention to treat population
Time Frame: Baseline
Population: Pediatric and Adult intent-to-treat (ITT) and per protocol (PP) populations. ITT population received at least one dose of study drug and one post-baseline assessment of the primary/secondary efficacy variables. PP population was participants that completed 12 months of treatment, had a valid assessment of the primary efficacy variable at Week 24.
Measure: Mean (Standard Deviation); unit: μg
Arm/Group | Pediatric Patients: Omalizumab + Budesonide and Formoterol | Pediatric Patients: Budesonide and Formoterol | Adult Patients: Omalizumab + Budesonide and Formoterol | Adult Patients: Budesonide and Formoterol
Number analyzed (Participants) | 16 | 17 | 40 | 39
μg
  ITT | 337.5 (95.74) | 270.6 (98.52) | 580.0 (201.53) | 533.3 (248.50)
  PP: number analyzed (Participants) | 11 | 12 | 32 | 33
  PP | 363.6 (80.90) | 250.0 (90.45) | 575.0 (201.61) | 533.3 (258.20)

2. Secondary Outcome: Number of Hospital Admissions Due to Asthma Exacerbation
Description: A hospital admission is defined as admissions to hospital involving a stay of at least 24 hours.
Time Frame: 12 month treatment duration
Population: Pediatric and Adult ITT population. ITT population received at least one dose of study drug and one post-baseline assessment of the primary/secondary efficacy variables.
Measure: Number; unit: hospital admissions
Arm/Group | Pediatric Patients: Omalizumab + Budesonide and Formoterol | Pediatric Patients: Budesonide and Formoterol | Adult Patients: Omalizumab + Budesonide and Formoterol | Adult Patients: Budesonide and Formoterol
Number analyzed (Participants) | 16 | 17 | 40 | 39
hospital admissions | 0 | 1 | 0 | 0

3. Secondary Outcome: Days Missed in School/Work Due to Asthma Exacerbation Episodes
Description: Participants /parent/legal guarding reported number of missed days of school or work at each study visit via diaries.
Time Frame: 12 month treatment duration
Population: as for outcome 2
Measure: Number; unit: days
Arm/Group | Pediatric Patients: Omalizumab + Budesonide and Formoterol | Pediatric Patients: Budesonide and Formoterol | Adult Patients: Omalizumab + Budesonide and Formoterol | Adult Patients: Budesonide and Formoterol
Number analyzed (Participants) | 16 | 17 | 40 | 39
days
  Missed school days | 2 | 3 | 1 | 0
  Missed work days | 0 | 1 | 0 | 1

4. Secondary Outcome: Control of Asthma Symptoms- Daytime Symptoms
Description: The clinical control of asthma was defined according to the following criteria (GINA 2012): 1-Daytime symptoms: none or less than twice a week 2-Limitations of daily activities: none 3-Nocturnal symptoms or awakening because of asthma: none 4-Need of relief or rescue medication: none or less than twice a week 5-Lung function (PEF or FEV1) without administration of bronchodilator: normal
Time Frame: 12 month treatment duration
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Pediatric Patients: Omalizumab + Budesonide and Formoterol | Pediatric Patients: Budesonide and Formoterol | Adult Patients: Omalizumab + Budesonide and Formoterol | Adult Patients: Budesonide and Formoterol
Number analyzed (Participants) | 16 | 17 | 40 | 39
percentage of participants | 62.5 | 70.6 | 82.5 | 71.8

5. Secondary Outcome: Control of Asthma Symptoms
Description: as for outcome 4
Time Frame: 12 month treatment duration
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Number of days
Arm/Group | Pediatric Patients: Omalizumab + Budesonide and Formoterol | Pediatric Patients: Budesonide and Formoterol | Adult Patients: Omalizumab + Budesonide and Formoterol | Adult Patients: Budesonide and Formoterol
Number analyzed (Participants) | 16 | 17 | 40 | 39
Number of days
  Wheezing: number analyzed (Participants) | 11 | 15 | 32 | 35
  Wheezing | 15.4 (23.43) | 21.1 (32.84) | 25.4 (28.89) | 29.0 (36.30)
  Night time cough: number analyzed (Participants) | 13 | 17 | 33 | 33
  Night time cough | 12.8 (7.75) | 20.8 (27.24) | 20.6 (22.09) | 32.3 (42.50)

6. Secondary Outcome: Control of Asthma Symptoms- Rescue Medication Use
Description: as for outcome 4
Time Frame: 12 month treatment duration
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Pediatric Patients: Omalizumab + Budesonide and Formoterol | Pediatric Patients: Budesonide and Formoterol | Adult Patients: Omalizumab + Budesonide and Formoterol | Adult Patients: Budesonide and Formoterol
Number analyzed (Participants) | 16 | 17 | 40 | 39
participants | 9 | 15 | 34 | 33

7. Secondary Outcome: Participants Requiring Oral Systemic Corticosteroids During the 12 Month Study Duration
Description: Number of days of concomitant medications use reported by participants at all visits via diaries.
Time Frame: 12 month treatment duration
Population: Number of patients requiring oral systemic corticosteroids within the ITT Pediatric and Adult population.
Measure: Mean (Standard Deviation); unit: Number of days
Groups:
- Adult Patients: Budesonide and Formoterol: Participants received budesonide + formoterol administered through an inhaler device.
Arm/Group | Pediatric Patients: Omalizumab + Budesonide and Formoterol | Pediatric Patients: Budesonide and Formoterol | Adult Patients: Omalizumab + Budesonide and Formoterol | Adult Patients: Budesonide and Formoterol
Number analyzed (Participants) | 3 | 2 | 5 | 9
Number of days | 7.3 (4.62) | 16.5 (19.09) | 28.0 (35.67) | 16.3 (17.35)

8. Secondary Outcome: Asthma Control Questionnaire (ACQ) at Baseline
Description: The Asthma Control Questionnaire (ACQ) has six questions to be answered by the participants, each with a 7 point scale (0-good control, 6-poor control), and one question where the actual pre-bronchodilator Forced expiratory volume in 1 second (FEV1) value expressed in % of predicted FEV1 was classified to scores from 0 (> 95% of predicted) to 6 (< 50% of predicted). The overall score is the average of the 7 questions; a minimum overall score of 0 = good control of asthma whereas a maximum overall score of 6 = poor control of asthma.
Time Frame: Baseline
Population: Number of participants with a baseline measurement within the ITT Pediatric and Adult population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pediatric Patients: Omalizumab + Budesonide and Formoterol | Pediatric Patients: Budesonide and Formoterol | Adult Patients: Omalizumab + Budesonide and Formoterol | Adult Patients: Budesonide and Formoterol
Number analyzed (Participants) | 15 | 17 | 40 | 39
scores on a scale | 3.3 (1.31) | 3.3 (1.26) | 3.6 (1.09) | 3.3 (1.35)

9. Secondary Outcome: Asthma Quality of Life Questionnaire (AQLQ) at Baseline
Description: The quality of life will be measured by the standardized version of the Asthma Quality of Life Questionnaire (AQLQ[S]) score for adults and the pediatric version of the AQLQ(S) for pediatric participants (PAQLQ[S]) . The AQLQ(S) and PAQLQ(S0 contain 4 domains (activity limitations, symptoms, emotional function, and environmental stimuli), with a total of 32 items; each item is measured in a 7-point Likert scale of 1 to 7 (1 = severe impairment, 7 = no impairment). All items are weighted equally. Mean score is calculated across all items within each domain and the overall score is the mean score of the 32 items.
Time Frame: Baseline
Population: Number of participants with a baseline measurement within the ITT Pediatric and Adult population.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pediatric Patients: Omalizumab + Budesonide and Formoterol | Pediatric Patients: Budesonide and Formoterol | Adult Patients: Omalizumab + Budesonide and Formoterol | Adult Patients: Budesonide and Formoterol
Number analyzed (Participants) | 15 | 17 | 40 | 39
scores on a scale
  Overall | 3.2 (1.21) | 3.4 (1.54) | 2.9 (1.04) | 3.4 (1.25)
  Symptoms domain | 3.2 (1.49) | 3.3 (1.48) | 2.8 (1.16) | 3.5 (1.37)
  Activity limitations domain | 3.2 (1.18) | 3.3 (1.47) | 3.2 (1.07) | 3.5 (1.25)
  Emotional functions domain | 3.2 (1.47) | 3.6 (1.76) | 2.5 (1.16) | 3.2 (1.49)
  Environmental stimuli domain | NA (NA) — Environment domain is non-existent for pediatric population. | NA (NA) — Environment domain is non-existent for pediatric population. | 2.7 (1.24) | 3.1 (1.47)

ADVERSE EVENTS:
Time Frame: Up to 12 months.
Arm/Group | Pediatric Patients: Omalizumab + Budesonide and Formoterol | Pediatric Patients: Budesonide and Formoterol | Adult Patients: Omalizumab + Budesonide and Formoterol | Adult Patients: Budesonide and Formoterol
Serious Adverse Events (participants affected / at risk) | 1/16 | 2/17 | 2/40 | 1/39
Other Adverse Events (participants affected / at risk) | 11/16 | 7/17 | 27/40 | 21/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pediatric Patients: Omalizumab + Budesonide and Formoterol (N=16) | Pediatric Patients: Budesonide and Formoterol (N=17) | Adult Patients: Omalizumab + Budesonide and Formoterol (N=40) | Adult Patients: Budesonide and Formoterol (N=39)
Food allergy (Immune system disorders) | 0 | 1 | 0 | 0
Maternal exposure during pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pelvic inflammatory disease (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Expired product administered (Product Issues) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pediatric Patients: Omalizumab + Budesonide and Formoterol (N=16) | Pediatric Patients: Budesonide and Formoterol (N=17) | Adult Patients: Omalizumab + Budesonide and Formoterol (N=40) | Adult Patients: Budesonide and Formoterol (N=39)
Increased hunger (Endocrine disorders) | 0 | 0 | 4 | 0
Burning in the eye (Eye disorders) | 0 | 0 | 1 | 2
Conjuntivitis - bacterial (Eye disorders) | 0 | 1 | 0 | 0
Pruritus - ocular (Eye disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain -localized (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Epigastric pain - food-related (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastroenteritis - acute (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 3 | 1
Hepatic steatosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Pyelonephritis - acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Adynamia (General disorders) | 1 | 0 | 1 | 0
Anxiety (General disorders) | 1 | 0 | 5 | 1
Asthenia (General disorders) | 1 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 1
Fever (General disorders) | 1 | 0 | 3 | 2
Pain (General disorders) | 0 | 0 | 2 | 1
Palpitations (General disorders) | 1 | 0 | 4 | 1
Tachycardia (General disorders) | 1 | 0 | 4 | 2
Diarrhea - Acute (Infections and infestations) | 1 | 0 | 0 | 0
External Otitis (Infections and infestations) | 1 | 0 | 0 | 0
Flu - common (Infections and infestations) | 0 | 0 | 0 | 3
flu-like symptoms (Infections and infestations) | 0 | 0 | 5 | 4
Influenza virus infection (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 2 | 1
Pharyngitis - Acute (Infections and infestations) | 1 | 0 | 1 | 1
Pharyngitis - bacterial (Infections and infestations) | 2 | 1 | 1 | 1
Pharyngotonsillitis (Infections and infestations) | 2 | 1 | 3 | 7
Rhinopharyngitis (Infections and infestations) | 2 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1
Sore throat (Infections and infestations) | 0 | 0 | 4 | 1
Tonsillitis - acute (Infections and infestations) | 0 | 0 | 1 | 2
Pruritus - injection site reaction (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Sea food allergy (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hands tremor (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Lower Limb cramp (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 3
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Muscle pain - localized (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Pain - leg (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Pain - localized (Musculoskeletal and connective tissue disorders) | 2 | 0 | 5 | 0
Tremor (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 1
Head trauma (Nervous system disorders) | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 2 | 3 | 5 | 3
Insomnia (Nervous system disorders) | 1 | 0 | 1 | 0
Lipothymia (Nervous system disorders) | 0 | 0 | 2 | 0
Allergic asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4 | 1
Cough - dry (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Cough - with sputum (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
CRUP syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Flu illness (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Nose bleeding (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Odinofagia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 5 | 0
Otorhinolaryngological examination (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Rhinitis - acute (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Rhinitis - allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 5 | 0
Rhinosinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1
Runny nose (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4 | 4
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5 | 3
Sputum (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5 | 2
Sputum increase (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Pruritus - allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.